CLINICAL TRIAL: NCT05496972
Title: Survey Assessment of Patient and Provider Impressions of Telemedicine in Radiation Oncology
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1063; NCI-2021-09908 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telemedicine Visits: Participants are asked to fill out a survey about their experience.
  Interventions: Behavioral: Survey Administration

INTERVENTIONS:
Behavioral: Survey Administration — Patients and providers complete survey over 10 minutes about their perspectives on the use of telemedicine

SUMMARY:
To understand more about the opinions of patients and health providers on the use of telemedicine in radiation oncology.

DETAILED DESCRIPTION:
Primary Objective:

To characterize patient and provider satisfaction with telemedicine in RO

Secondary Objective:

* To provide evidence for or against the use of telemedicine in radiation oncology (RO)
* To assess the feasibility of and value added by telemedicine in RO
* To describe barriers and facilitators to telemedicine in RO
* To identify preferred use cases for telemedicine in RO

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they are aged 18 or older and have undergone at least 1 telemedicine encounter (video visit) with the radiation oncology department at MD Anderson or its affiliates within 2 months from the initiation of the study (and prospectively as the study enrolls). This would include weekly see visits, follow-up visits, or consultations
* English speaking
* Access to email and internet to complete the survey
* Attending physicians in the radiation oncology department who have utilized telemedicine will be contacted to fill out surveys reflecting their experience

Exclusion Criteria:

• Protected populations such as adults unable to consent, pregnant women, prisoners, and individuals who are not yet adults will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction survey with telemedicine in radiation oncology (RO) | through study completion and average of one year.
  Sensitivity analyses will be performed with those rating 9 or higher or less than 9, and for those who "agree" or "strongly agree" with whether they are satisfied with telemedicine compared to those who give other answers.
Provider satisfaction survey with telemedicine in radiation oncology (RO) | through study completion and average of one year.
  Sensitivity analyses will be performed with those rating 9 or higher or less than 9, and for those who "agree" or "strongly agree" with whether they are satisfied with telemedicine compared to those who give other answers.

CONTACTS AND LOCATIONS:
Overall Officials: Chenyang Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org